CLINICAL TRIAL: NCT06290206
Title: PREVENT: Practice-based Approaches to Promote HPV Vaccination in the Safety Net - BootCamp Translation
Brief Title: PREVENT HPV-Related Cancers - BootCamp Translation
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Kaiser Permanente (Other); University of Arizona (Other); Sea Mar Community Health Centers (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCI161649-1; 1R01CA279973-01 (NIH); DSS_10065815 (Other: University of Utah, Document Summary Sheet (DSS) Number)
Record Dates: First submitted 2024-02-04; First posted 2024-03-04 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: HPV Vaccination; Vaccine; Uptake; Vaccination; Series Completion
Keywords: Humans; Adolescent; Child; Male; Female; Caregivers; Parents; Hispanic or Latino; Rural Population; Health Personnel; United States; Vaccination; Papillomavirus Vaccines; Papillomavirus Vaccines / administration & dosage; Human Papillomavirus Viruses; Papillomavirus Infections; Papillomavirus Infections / prevention & control; Cancer / prevention & control; Incidence; Text Messaging; Reminder Systems / instrumentation; Social Norms; Vaccination Refusal; Health Knowledge, Attitudes, Practice; Health Promotion / methods; Motivation; Communication; Patient Acceptance of Health Care; Parents / education; Religion; Religiosity; Stakeholder Participation; Participatory Approach; Qualitative Research; Quantitative Research; Randomized Control Trial; Surveys and Questionnaires
MeSH Terms: conditions — Papillomavirus Infections; Neoplasms; Vaccination Refusal; Behavior; Communication; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- English Language Session and Messaging (Experimental): The in-person or live Zoom presentation in English will consist of an expert presentation about the research on the safety and effectiveness of the HPV vaccine and social norms about vaccination. In this session, participants will receive up-to-date evidence on effective messaging by clinicians (e.g., using presumptive statements, bundling HPV vaccine recommendations with recommendations for other vaccines) in addition to novel formats for educational messages (e.g., digital videos, narratives).
  Participants in the English-language text message group will provide iterative feedback to the research team on HPV vaccination messages over a 3-month period.
  Interventions: Behavioral: PREVENT - BCT
- Spanish Language Session and Messaging (Experimental): The in-person or live Zoom presentation in Spanish will consist of an expert presentation about the research on the safety and effectiveness of the HPV vaccine and social norms about vaccination. In this session, participants will receive up-to-date evidence on effective messaging by clinicians (e.g., using presumptive statements, bundling HPV vaccine recommendations with recommendations for other vaccines) in addition to novel formats for educational messages (e.g., digital videos, narratives).
  Participants in the Spanish-language text message group will provide iterative feedback to the research team on HPV vaccination messages over a 3-month period.
  Interventions: Behavioral: PREVENT - BCT

INTERVENTIONS:
Behavioral: PREVENT - BCT — Bootcamp Translation (BCT), a method for engaging diverse stakeholders in a consensus-building process, has been used by this research team to actively develop and adapt study interventions. It uses an iterative, flexible schedule of face-to-face meetings combined with short, focused teleconferences. BCT emphasizes no wrong answers and no hierarchy of expertise. The process requires up to nine (9) hours of participant time over 3-6 months. Participants will be surveyed before and after the in-person session to assess learning outcomes and capture basic sociodemographic information.
  The BCT process will define the format (mode and frequency) and content of messages to promote vaccine series completion. Auto and Auto-Plus intervention arms may use some of the same components (automated calls, live calls, text messages, emails, and mailings).

SUMMARY:
This study will serve as one of the first to develop and test the effectiveness of strategies to promote HPV vaccination among diverse rural parents and caregivers of children ages 9-17 years in the Mountain West. Once implemented into practice, this intervention could significantly reduce disparities in the burden of HPV-associated cancers among rural populations in the United States.

The proposed study will determine the components of clinic-based outreach to increase vaccination rates for HPV at four community clinics in rural counties in Washington. This study is a boot camp translation to tailor messaging based on patient and provider input.

This study will refine intervention components and messages to increase HPV vaccination among rural children and adolescents (C/A). The research team will use a validated patient-engaged approach for parents/caregivers (P/Cs), Bootcamp Translation (BCT), with separate sessions conducted in English and Spanish.

DETAILED DESCRIPTION:
The PREVENT BootCamp Translation (BCT) study will determine the components and messages of reminders to encourage parents to obtain an HPV vaccine for their age-eligible children and adolescents (C/A)

This study will design format and content of an intervention to promote adolescent HPV vaccine coverage that will consider unique information needs of diverse rural parents/caregivers. The study team will use BCT to develop locally relevant intervention materials (e.g., reminder phone scripts for automated calls, text messages, and patient portal messages for P/C). Targeted promotional materials for HPV vaccination are available in Spanish and could be translated into other languages, as needed. Newly designed messages and materials will seek to counter anti-vaccination sentiment by leveraging cancer prevention, vaccine effectiveness, and vaccine safety messages. BCT methods will provide the framework to tailor HPV vaccination messages for rural and Hispanic IMW P/C.

Bootcamp Translation (BCT), a method for engaging diverse stakeholders in a consensus-building process, has been used by this research team to actively develop and adapt study interventions. It uses an iterative, flexible schedule of face-to-face meetings combined with short, focused teleconferences in a process that addresses 2 questions: "What do we need to say in our message to the community (newly HPV vaccine-eligible adolescents and adolescents who have not completed the HPV vaccination series)?" and "How do we deliver that message to our community?" BCT emphasizes no wrong answers and no hierarchy of expertise. The process requires up to nine (9) hours of participant time over 3-6 months. Participants will be surveyed before and after the in-person session to assess learning outcomes and capture basic sociodemographic information.

With Sea Mar's project manager and/or Sea Mar's designated team member(s), this study will recruit P/C (i.e., participants) for BCT sessions by generating a list of potential P/C of patients across 4 clinics. This study will recruit 6 participants from each clinic (24 total): 12 whose preferred language is English and 12 whose preferred language is Spanish. About two Sea Mar staff members will participate in BCT.

Two parallel sessions will be conducted, one in English and one in Spanish, with approximately 12 study participants per session. The in-person or live Zoom presentation will consist of an expert presentation, and/or subject matter experts. They will share research on the safety and effectiveness of the HPV vaccine and social norms about vaccination. They will educate participants about the six different types of cancers that are prevented by the HPV vaccine among women and men in the United States. The study Investigators and/or subject matter experts to whom they delegate this responsibility will also present up-to-date evidence on effective messaging by clinicians (e.g., using presumptive statements, bundling HPV vaccine recommendations with recommendations for other vaccines) as well as novel formats for educational messages (e.g., digital videos, narratives).

Participants will be assigned to a Spanish-language or English-language text message group, as appropriate, to provide iterative feedback to the research team on HPV vaccination messages over a 3-month period. Clinical partners in rural communities emphasized the high prevalence of mobile phone use among the parents/caregivers in their communities for seeking and sharing health information, and nationally 95% of adults ages 18-49 have a smartphone, including the majority of Hispanics (85%) and rural residents (80%). Further, obtaining feedback from P/C about the suitability of HPV vaccine messages through text messaging will facilitate more specific and tailored feedback from participants, increase accessibility for individuals who may have limited access to meet in person, and provide an opportunity where individuals may feel more comfortable sharing their opinions and perceptions than they would during a face-to-face or synchronous online experience. Text messages will emphasize individual involvement and personal meaning to enhance retention and promote engagement. Text messages between study staff and BCT participants will occur through the text messaging Twillio, which the research team has previously used to pilot HPV vaccine reminders. Text messages will be designed to elicit feedback on the HPV vaccination messages (which are suitable for girls vs. boys, English vs. Spanish speaking parents/caregivers) that are developed during the Bootcamp sessions, on reminder scripts (i.e., automated call scripts, text messages, patient portal messages), and on key intervention components (e.g., reminder type, number, sequence). The text messages will occur two times per week. This process can be automated using the text-messaging tool Twillio. Each text will ask participants to provide their feedback via text response. Messages will be pilot tested.

Because the BCT process is interactive and iterative, recording and transcribing sessions is often impractical. Instead, field notes will be taken by the study team in English and/or Spanish during each session and shared during weekly meetings of the project team. Reminder materials tailored through BCT and proposed protocols for the intervention will be reviewed by members of the IMW HPV Vaccination Coalition and tested in a later study. Following BCT, the research team will finalize the trial protocol, including procedures for the Auto and the Auto-Plus arms of the intervention, and the study team will finalize methods for data coordination, management, and ongoing monitoring. Because the goal of this study is to craft materials and messages that are motivating for English- and Spanish-speakers, this study does not anticipate directly translating materials from English to Spanish. Instead, the research team will rely on BCT and native speakers to craft messages from the ground up; this approach was successful in prior research. This study aims for a broad scale-up, all English and Spanish materials will be reviewed by the Sea Mar marketing and communications office for appropriateness and equivalency.

ELIGIBILITY:
Inclusion Criteria:

1. Parents/Caregivers (P/C) of children/adolescents (C/A) ages 9-17 years of age (i.e., age-eligible for HPV vaccination);
2. P/C with active clinic patients (i.e., have been seen in the clinic in the last 12 months); and
3. P/C who speak either English or Spanish.

Exclusion Criteria:

1. P/C of C/A with previous excluding HPV vaccination history (e.g., completed vaccination, or not due);
2. P/C of C/A with clinical conditions that influence the CDC HPV vaccination recommendations (e.g., pregnancy);
3. P/C of C/A with other factors that would influence CDC HPV recommendations; and
4. P/C that does not speak Spanish or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Kepka, PhD, MPH, Principal Investigator — Huntsman Cancer Institute/ University of Utah; Medical Director, MD, Study Chair — Sea Mar
Locations (1):
- Sea Mar Community Health Centers, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
A plan for sharing IDP that maintains participant anonymity has not yet been developed.

REFERENCES:
- [Background] Saslow D, Andrews KS, Manassaram-Baptiste D, Loomer L, Lam KE, Fisher-Borne M, Smith RA, Fontham ET; American Cancer Society Guideline Development Group. Human papillomavirus vaccination guideline update: American Cancer Society guideline endorsement. CA Cancer J Clin. 2016 Sep;66(5):375-85. doi: 10.3322/caac.21355. Epub 2016 Jul 19. PMID 27434803
- [Background] Tabak RG, Duggan K, Smith C, Aisaka K, Moreland-Russell S, Brownson RC. Assessing Capacity for Sustainability of Effective Programs and Policies in Local Health Departments. J Public Health Manag Pract. 2016 Mar-Apr;22(2):129-37. doi: 10.1097/PHH.0000000000000254. PMID 25946700
- [Background] Brownson RC, Reis RS, Allen P, Duggan K, Fields R, Stamatakis KA, Erwin PC. Understanding administrative evidence-based practices: findings from a survey of local health department leaders. Am J Prev Med. 2014 Jan;46(1):49-57. doi: 10.1016/j.amepre.2013.08.013. PMID 24355671
- [Background] Shea CM, Jacobs SR, Esserman DA, Bruce K, Weiner BJ. Organizational readiness for implementing change: a psychometric assessment of a new measure. Implement Sci. 2014 Jan 10;9:7. doi: 10.1186/1748-5908-9-7. PMID 24410955
- [Background] Wutich A, Bernard HR. Sharing qualitative data & analysis. With whom and how widely?: A response to 'Promises and pitfalls of data sharing in qualitative research'. Soc Sci Med. 2016 Nov;169:199-200. doi: 10.1016/j.socscimed.2016.09.041. Epub 2016 Sep 30. No abstract available. PMID 27720554
- [Background] Patton MQ. Qualitative research and evaluation methods. Thousand Oaks, CA: Sage Publications, Inc.; 2002
- [Background] Malterud K, Siersma VD, Guassora AD. Sample Size in Qualitative Interview Studies: Guided by Information Power. Qual Health Res. 2016 Nov;26(13):1753-1760. doi: 10.1177/1049732315617444. Epub 2016 Jul 10. PMID 26613970
- [Background] Silverman D. Qualitative Research: A practical handbook. Thousand Oaks, CA: Sage Publications, Inc.; 2010.
- [Background] Nonzee NJ, Baldwin SB, Cui Y, Singhal R. Disparities in parental human papillomavirus (HPV) vaccine awareness and uptake among adolescents. Vaccine. 2018 Feb 28;36(10):1243-1247. doi: 10.1016/j.vaccine.2017.08.046. Epub 2017 Sep 28. PMID 28967520
- [Background] Choi Y, Eworuke E, Segal R. What explains the different rates of human papillomavirus vaccination among adolescent males and females in the United States? Papillomavirus Res. 2016 Dec;2:46-51. doi: 10.1016/j.pvr.2016.02.001. Epub 2016 Mar 4. PMID 29074185
- [Background] Warner EL, Ding Q, Pappas L, Bodson J, Fowler B, Mooney R, Kirchhoff AC, Kepka D. Health Care Providers' Knowledge of HPV Vaccination, Barriers, and Strategies in a State With Low HPV Vaccine Receipt: Mixed-Methods Study. JMIR Cancer. 2017 Aug 11;3(2):e12. doi: 10.2196/cancer.7345. PMID 28801303
- [Background] Garcia AA, Zuniga JA, Lagon C. A Personal Touch: The Most Important Strategy for Recruiting Latino Research Participants. J Transcult Nurs. 2017 Jul;28(4):342-347. doi: 10.1177/1043659616644958. Epub 2016 Apr 25. PMID 27114390
- [Background] Kim SY, Chen S, Hou Y, Zeiders KH, Calzada EJ. Parental socialization profiles in Mexican-origin families: Considering cultural socialization and general parenting practices. Cultur Divers Ethnic Minor Psychol. 2019 Jul;25(3):439-450. doi: 10.1037/cdp0000234. Epub 2018 Nov 1. PMID 30382707
- [Background] Coronado GD, Petrik A, Spofford M, Talbot J, Do HH, Sanchez J, Kapka T, Taylor V. Perceptions of under and overutilization of cervical cancer screening services at Latino-serving community health centers. J Community Health. 2013 Oct;38(5):915-8. doi: 10.1007/s10900-013-9701-1. PMID 23728821
- [Background] Jackson ML, Henrikson NB, Grossman DC. Evaluating Washington State's immunization information system as a research tool. Acad Pediatr. 2014 Jan-Feb;14(1):71-6. doi: 10.1016/j.acap.2013.10.002. PMID 24369871
- [Background] Maneesriwongul W, Dixon JK. Instrument translation process: a methods review. J Adv Nurs. 2004 Oct;48(2):175-86. doi: 10.1111/j.1365-2648.2004.03185.x. PMID 15369498
- [Background] Centers for Disease Control and Prevention. Human Papillomavirus (HPV). Educational Materials. Available from: https://www.cdc.gov/hpv/hcp/educational-materials.html.
- [Background] Moorhead SA, Hazlett DE, Harrison L, Carroll JK, Irwin A, Hoving C. A new dimension of health care: systematic review of the uses, benefits, and limitations of social media for health communication. J Med Internet Res. 2013 Apr 23;15(4):e85. doi: 10.2196/jmir.1933. PMID 23615206
- [Background] Pew Research Center. Mobile Fact Sheet. Available from: https://www.pewresearch.org/internet/fact-sheet/mobile/
- [Background] Tiro JA, Sanders JM, Pruitt SL, Stevens CF, Skinner CS, Bishop WP, Fuller S, Persaud D. Promoting HPV Vaccination in Safety-Net Clinics: A Randomized Trial. Pediatrics. 2015 Nov;136(5):850-9. doi: 10.1542/peds.2015-1563. Epub 2015 Oct 19. PMID 26482674
- [Background] Calo WA, Gilkey MB, Malo TL, Robichaud M, Brewer NT. A content analysis of HPV vaccination messages available online. Vaccine. 2018 Nov 26;36(49):7525-7529. doi: 10.1016/j.vaccine.2018.10.053. Epub 2018 Oct 23. PMID 30366803
- [Background] undefined
- [Background] Nan X, Madden K, Richards A, Holt C, Wang MQ, Tracy K. Message Framing, Perceived Susceptibility, and Intentions to Vaccinate Children Against HPV Among African American Parents. Health Commun. 2016 Jul;31(7):798-805. doi: 10.1080/10410236.2015.1005280. Epub 2015 Dec 8. PMID 26646190
- [Background] Mroz S, Zhang X, Williams M, Conlon A, LoConte NK. Working to Increase Vaccination for Human Papillomavirus: A Survey of Wisconsin Stakeholders, 2015. Prev Chronic Dis. 2017 Sep 28;14:E85. doi: 10.5888/pcd14.160610. PMID 28957034
- [Background] Thompson JH, Davis MM, Michaels L, Rivelli JS, Castillo ML, Younger BM, Castro M, Reich SL, Coronado GD. Developing Patient-Refined Messaging for a Mailed Colorectal Cancer Screening Program in a Latino-Based Community Health Center. J Am Board Fam Med. 2019 May-Jun;32(3):307-317. doi: 10.3122/jabfm.2019.03.180026. PMID 31068395
- [Background] National Heart Lung and Blood Institute. Research dissemination and implementation (R18) grants2011 01/09/2012. Available from: http://www.nhlbi.nih.gov/funding/policies/dissemination&implementationR18.htm.
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Estabrooks PA, Vogt TM. Evaluating the impact of health promotion programs: using the RE-AIM framework to form summary measures for decision making involving complex issues. Health Educ Res. 2006 Oct;21(5):688-94. doi: 10.1093/her/cyl081. Epub 2006 Aug 31. PMID 16945984
- [Background] Glasgow RE, Wagner EH, Schaefer J, Mahoney LD, Reid RJ, Greene SM. Development and validation of the Patient Assessment of Chronic Illness Care (PACIC). Med Care. 2005 May;43(5):436-44. doi: 10.1097/01.mlr.0000160375.47920.8c. PMID 15838407
- [Background] Glasgow RE, Ory MG, Klesges LM, Cifuentes M, Fernald DH, Green LA. Practical and relevant self-report measures of patient health behaviors for primary care research. Ann Fam Med. 2005 Jan-Feb;3(1):73-81. doi: 10.1370/afm.261. PMID 15671195
- [Background] Glasgow RE, Klesges LM, Dzewaltowski DA, Bull SS, Estabrooks P. The future of health behavior change research: what is needed to improve translation of research into health promotion practice? Ann Behav Med. 2004 Feb;27(1):3-12. doi: 10.1207/s15324796abm2701_2. PMID 14979858
- [Background] National Cancer Institute. How do RE-AIM elements relate to planning? 2011 01/05/2012. Available from: http://cancercontrol.cancer.gov/IS/reaim/faq.html#define.
- [Background] Glasgow RE. RE-AIMing research for application: ways to improve evidence for family medicine. J Am Board Fam Med. 2006 Jan-Feb;19(1):11-9. doi: 10.3122/jabfm.19.1.11. PMID 16492000
- [Background] Thompson JH, Davis MM, Leo MC, Schneider JL, Smith DH, Petrik AF, Castillo M, Younger B, Coronado GD. Participatory Research to Advance Colon Cancer Prevention (PROMPT): Study protocol for a pragmatic trial. Contemp Clin Trials. 2018 Apr;67:11-15. doi: 10.1016/j.cct.2018.02.001. Epub 2018 Feb 9. PMID 29408304
- [Background] Westfall JM, Zittleman L, Sutter C, Emsermann CB, Staton EW, Van Vorst R, Dickinson LM; Community Advisory Council. Testing to prevent colon cancer: results from a rural community intervention. Ann Fam Med. 2013 Nov-Dec;11(6):500-7. doi: 10.1370/afm.1582. PMID 24218373
- [Background] Norman N, Bennett C, Cowart S, Felzien M, Flores M, Flores R, Haynes C, Hernandez M, Rodriquez MP, Sanchez N, Sanchez S, Winkelman K, Winkelman S, Zittleman L, Westfall JM. Boot camp translation: a method for building a community of solution. J Am Board Fam Med. 2013 May-Jun;26(3):254-63. doi: 10.3122/jabfm.2013.03.120253. PMID 23657693
- [Background] Satcher, D. (2005). Methods in community-based participatory research for health. John Wiley & Sons.
- [Background] SeaMar Community Health Centers (Clinica de la Comunidad). Report to the Community2018 02/26/2019. Available from: https://seamar.org/seamar-downloads/Annual-Report2018.pdf
- [Background] Coronado GD, Golovaty I, Longton G, Levy L, Jimenez R. Effectiveness of a clinic-based colorectal cancer screening promotion program for underserved Hispanics. Cancer. 2011 Apr 15;117(8):1745-54. doi: 10.1002/cncr.25730. Epub 2010 Nov 8. PMID 21472722
- [Background] Edwards BK, Ward E, Kohler BA, Eheman C, Zauber AG, Anderson RN, Jemal A, Schymura MJ, Lansdorp-Vogelaar I, Seeff LC, van Ballegooijen M, Goede SL, Ries LA. Annual report to the nation on the status of cancer, 1975-2006, featuring colorectal cancer trends and impact of interventions (risk factors, screening, and treatment) to reduce future rates. Cancer. 2010 Feb 1;116(3):544-73. doi: 10.1002/cncr.24760. PMID 19998273
- [Background] Parker E, Margolis LH, Eng E, Henriquez-Roldan C. Assessing the capacity of health departments to engage in community-based participatory public health. Am J Public Health. 2003 Mar;93(3):472-6. doi: 10.2105/ajph.93.3.472. PMID 12604498
- [Background] Thompson B, Coronado G, Snipes SA, Puschel K. Methodologic advances and ongoing challenges in designing community-based health promotion programs. Annu Rev Public Health. 2003;24:315-40. doi: 10.1146/annurev.publhealth.24.100901.140819. Epub 2001 Nov 6. PMID 12471272
- [Background] University of Washington. Developing and Sustaining Community Based Participatory Research Partnerships: A Skill Building Curriculum2012 04/21/2012 Available from: http://depts.washington.edu/ccph/cbpr/u1/u11.php.
- [Background] University of Washington School of Public Health and Community Medicine. Community-based research principles. Available from: http://sphcm.washington.edu/research/community.htm.
- [Background] Byrd TL, Wilson KM, Smith JL, Coronado G, Vernon SW, Fernandez-Esquer ME, Thompson B, Ortiz M, Lairson D, Fernandez ME. AMIGAS: a multicity, multicomponent cervical cancer prevention trial among Mexican American women. Cancer. 2013 Apr 1;119(7):1365-72. doi: 10.1002/cncr.27926. Epub 2012 Dec 21. PMID 23280399
- [Background] Thompson B, Carosso EA, Jhingan E, Wang L, Holte SE, Byrd TL, Benavides MC, Lopez C, Martinez-Gutierrez J, Ibarra G, Gonzalez VJ, Gonzalez NE, Duggan CR. Results of a randomized controlled trial to increase cervical cancer screening among rural Latinas. Cancer. 2017 Feb 15;123(4):666-674. doi: 10.1002/cncr.30399. Epub 2016 Oct 27. PMID 27787893
- [Background] Duggan C, Coronado G, Martinez J, Byrd TL, Carosso E, Lopez C, Benavides M, Thompson B. Cervical cancer screening and adherence to follow-up among Hispanic women study protocol: a randomized controlled trial to increase the uptake of cervical cancer screening in Hispanic women. BMC Cancer. 2012 May 6;12:170. doi: 10.1186/1471-2407-12-170. PMID 22559251
- [Background] Coronado GD, Rivelli JS, Fuoco MJ, Vollmer WM, Petrik AF, Keast E, Barker S, Topalanchik E, Jimenez R. Effect of Reminding Patients to Complete Fecal Immunochemical Testing: A Comparative Effectiveness Study of Automated and Live Approaches. J Gen Intern Med. 2018 Jan;33(1):72-78. doi: 10.1007/s11606-017-4184-x. Epub 2017 Oct 10. PMID 29019046
- [Background] Coronado GD, Burdick T, Petrik A, Kapka T, Retecki S, Green B. Using an Automated Data-driven, EHR-Embedded Program for Mailing FIT kits: Lessons from the STOP CRC Pilot Study. J Gen Pract (Los Angel). 2014 Jan 5;2:1000141. doi: 10.4172/2329-9126.1000141. PMID 25411657
- [Background] Kepka DL, Ulrich AK, Coronado GD. Low knowledge of the three-dose HPV vaccine series among mothers of rural Hispanic adolescents. J Health Care Poor Underserved. 2012 May;23(2):626-35. doi: 10.1353/hpu.2012.0040. PMID 22643612
- [Background] Kepka DL, Coronado GD, Rodriguez HP, Thompson B. Development of a radionovela to promote HPV vaccine awareness and knowledge among Latino parents. Public Health Rep. 2012 Jan-Feb;127(1):130-8. doi: 10.1177/003335491212700118. No abstract available. PMID 22298937
- [Background] Ayres S, Gee A, Kim S, Hashibe M, Praag A, Kaiser D, Chang CP, Brandt HM, Kepka D. Human Papillomavirus Vaccination Knowledge, Barriers, and Recommendations Among Healthcare Provider Groups in the Western United States. J Cancer Educ. 2022 Dec;37(6):1816-1823. doi: 10.1007/s13187-021-02047-6. Epub 2021 Jul 8. PMID 34236651
- [Background] Brandt HM, Kepka D, Kirchhoff AC, Daniel CL, Bhatt NS. Human papillomavirus (HPV) vaccination is cancer prevention for childhood cancer survivors. Cancer. 2022 Jan 15;128(2):237-239. doi: 10.1002/cncr.33920. Epub 2021 Oct 4. PMID 34606629
- [Background] Kepka D, Christini K, McGough E, Wagner A, Del Fiol G, Gibson B, Ayres S, Brandt HM, Mann S, Petrik AF, Coronado GD. Successful Multi-Level HPV Vaccination Intervention at a Rural Healthcare Center in the Era of COVID-19. Front Digit Health. 2021 Aug 19;3:719138. doi: 10.3389/fdgth.2021.719138. eCollection 2021. PMID 34713184
- [Background] Kepka D, Ding Q, Bodson J, Warner EL, Mooney K. Latino Parents' Awareness and Receipt of the HPV Vaccine for Sons and Daughters in a State with Low Three-Dose Completion. J Cancer Educ. 2015 Dec;30(4):808-12. doi: 10.1007/s13187-014-0781-0. PMID 25572463
- [Background] Warner EL, Lai D, Carbajal-Salisbury S, Garza L, Bodson J, Mooney K, Kepka D. Latino Parents' Perceptions of the HPV Vaccine for Sons and Daughters. J Community Health. 2015 Jun;40(3):387-94. doi: 10.1007/s10900-014-9949-0. PMID 25269400
- [Background] Kepka D, Warner EL, Kinney AY, Spigarelli MG, Mooney K. Low human papillomavirus (HPV) vaccine knowledge among Latino parents in Utah. J Immigr Minor Health. 2015 Feb;17(1):125-31. doi: 10.1007/s10903-014-0003-1. PMID 24609357
- [Background] Warner EL, Ding Q, Pappas LM, Henry K, Kepka D. White, affluent, educated parents are least likely to choose HPV vaccination for their children: a cross-sectional study of the National Immunization Study - teen. BMC Pediatr. 2017 Dec 1;17(1):200. doi: 10.1186/s12887-017-0953-2. PMID 29191180
- [Background] Islam JY, Gruber JF, Kepka D, Kunwar M, Smith SB, Rothholz MC, Brewer NT, Smith JS. Pharmacist insights into adolescent human papillomavirus vaccination provision in the United States. Hum Vaccin Immunother. 2019;15(7-8):1839-1850. doi: 10.1080/21645515.2018.1556077. Epub 2019 Feb 6. PMID 30550369
- [Background] Elam-Evans LD, Yankey D, Singleton JA, Sterrett N, Markowitz LE, Williams CL, Fredua B, McNamara L, Stokley S. National, Regional, State, and Selected Local Area Vaccination Coverage Among Adolescents Aged 13-17 Years - United States, 2019. MMWR Morb Mortal Wkly Rep. 2020 Aug 21;69(33):1109-1116. doi: 10.15585/mmwr.mm6933a1. PMID 32817598
- [Background] Vogelaar I, van Ballegooijen M, Schrag D, Boer R, Winawer SJ, Habbema JD, Zauber AG. How much can current interventions reduce colorectal cancer mortality in the U.S.? Mortality projections for scenarios of risk-factor modification, screening, and treatment. Cancer. 2006 Oct 1;107(7):1624-33. doi: 10.1002/cncr.22115. PMID 16933324
- [Background] Hopfer S, Garcia S, Duong HT, Russo JA, Tanjasiri SP. A Narrative Engagement Framework to Understand HPV Vaccination Among Latina and Vietnamese Women in a Planned Parenthood Setting. Health Educ Behav. 2017 Oct;44(5):738-747. doi: 10.1177/1090198117728761. Epub 2017 Aug 30. PMID 28854812
- [Background] Szilagyi PG, Humiston SG, Gallivan S, Albertin C, Sandler M, Blumkin A. Effectiveness of a citywide patient immunization navigator program on improving adolescent immunizations and preventive care visit rates. Arch Pediatr Adolesc Med. 2011 Jun;165(6):547-53. doi: 10.1001/archpediatrics.2011.73. PMID 21646588
- [Background] Vanderpool RC, Stradtman LR, Brandt HM. Policy opportunities to increase HPV vaccination in rural communities. Hum Vaccin Immunother. 2019;15(7-8):1527-1532. doi: 10.1080/21645515.2018.1553475. Epub 2019 Jan 4. PMID 30608894
- [Background] Brandt HM, Pierce JY, Crary A. Increasing HPV vaccination through policy for public health benefit. Hum Vaccin Immunother. 2016 Jun 2;12(6):1623-5. doi: 10.1080/21645515.2015.1122145. Epub 2015 Dec 15. PMID 26669416
- [Background] Khuwaja SS, Peck JL. Increasing HPV Vaccination Rates Using Text Reminders: An Integrative Review of the Literature. J Pediatr Health Care. 2022 Jul-Aug;36(4):310-320. doi: 10.1016/j.pedhc.2022.02.001. Epub 2022 Mar 11. PMID 35288016
- [Background] Francis DB, Cates JR, Wagner KPG, Zola T, Fitter JE, Coyne-Beasley T. Communication technologies to improve HPV vaccination initiation and completion: A systematic review. Patient Educ Couns. 2017 Jul;100(7):1280-1286. doi: 10.1016/j.pec.2017.02.004. Epub 2017 Feb 6. PMID 28209248
- [Background] Hou SI, Fernandez ME, Parcel GS. Development of a cervical cancer educational program for Chinese women using intervention mapping. Health Promot Pract. 2004 Jan;5(1):80-7. doi: 10.1177/1524839903257311. PMID 14965438
- [Background] Byrd TL, Wilson KM, Smith JL, Heckert A, Orians CE, Vernon SW, Fernandez-Esquer ME, Fernandez ME. Using intervention mapping as a participatory strategy: development of a cervical cancer screening intervention for Hispanic women. Health Educ Behav. 2012 Oct;39(5):603-11. doi: 10.1177/1090198111426452. Epub 2012 Mar 1. PMID 22388451
- [Background] Fernandez ME, Gonzales A, Tortolero-Luna G, Partida S, Bartholomew LK. Using intervention mapping to develop a breast and cervical cancer screening program for Hispanic farmworkers: Cultivando La Salud. Health Promot Pract. 2005 Oct;6(4):394-404. doi: 10.1177/1524839905278810. PMID 16210681
- [Background] Warner EL, Fowler B, Martel L, Kepka D. Improving HPV Vaccination Through a Diverse Multi-state Coalition. J Community Health. 2017 Oct;42(5):911-920. doi: 10.1007/s10900-017-0334-7. PMID 28393294
- [Background] Bartholomew LK, Parcel GS, Kok G. Intervention mapping: a process for developing theory- and evidence-based health education programs. Health Educ Behav. 1998 Oct;25(5):545-63. doi: 10.1177/109019819802500502. PMID 9768376
- [Background] Paskett ED, Krok-Schoen JL, Pennell ML, Tatum CM, Reiter PL, Peng J, Bernardo BM, Weier RC, Richardson MS, Katz ML. Results of a Multilevel Intervention Trial to Increase Human Papillomavirus (HPV) Vaccine Uptake among Adolescent Girls. Cancer Epidemiol Biomarkers Prev. 2016 Apr;25(4):593-602. doi: 10.1158/1055-9965.EPI-15-1243. PMID 27196093
- [Background] Fridman A, Gershon R, Gneezy A. COVID-19 and vaccine hesitancy: A longitudinal study. PLoS One. 2021 Apr 16;16(4):e0250123. doi: 10.1371/journal.pone.0250123. eCollection 2021. PMID 33861765
- [Background] Santibanez TA, Singleton JA, Santibanez SS, Wortley P, Bell BP. Socio-demographic differences in opinions about 2009 pandemic influenza A (H1N1) and seasonal influenza vaccination and disease among adults during the 2009-2010 influenza season. Influenza Other Respir Viruses. 2013 May;7(3):383-92. doi: 10.1111/j.1750-2659.2012.00374.x. Epub 2012 May 9. PMID 22568588
- [Background] Arda B, Durusoy R, Yamazhan T, Sipahi OR, Tasbakan M, Pullukcu H, Erdem E, Ulusoy S. Did the pandemic have an impact on influenza vaccination attitude? A survey among health care workers. BMC Infect Dis. 2011 Apr 7;11:87. doi: 10.1186/1471-2334-11-87. PMID 21473763
- [Background] Halperin BA, MacKinnon-Cameron D, McNeil S, Kalil J, Halperin SA. Maintaining the momentum: key factors influencing acceptance of influenza vaccination among pregnant women following the H1N1 pandemic. Hum Vaccin Immunother. 2014;10(12):3629-41. doi: 10.4161/21645515.2014.980684. PMID 25668670
- [Background] Quinn SC, Parmer J, Freimuth VS, Hilyard KM, Musa D, Kim KH. Exploring communication, trust in government, and vaccination intention later in the 2009 H1N1 pandemic: results of a national survey. Biosecur Bioterror. 2013 Jun;11(2):96-106. doi: 10.1089/bsp.2012.0048. Epub 2013 Apr 25. PMID 23617721
- [Background] Meyer AF, Borkovskiy NL, Brickley JL, Chaudhry R, Franqueira A, Furst JW, Hinsch DM, McDonah MR, Myers JF, Petersen RE, Finney Rutten LJ, Wilson PM, Jacobson RM. Impact of Electronic Point-of-Care Prompts on Human Papillomavirus Vaccine Uptake in Retail Clinics. Am J Prev Med. 2018 Dec;55(6):822-829. doi: 10.1016/j.amepre.2018.06.027. Epub 2018 Oct 19. PMID 30344033
- [Background] Henrikson NB, Zhu W, Baba L, Nguyen M, Berthoud H, Gundersen G, Hofstetter AM. Outreach and Reminders to Improve Human Papillomavirus Vaccination in an Integrated Primary Care System. Clin Pediatr (Phila). 2018 Nov;57(13):1523-1531. doi: 10.1177/0009922818787868. Epub 2018 Jul 13. PMID 30003794
- [Background] Larson HJ, Clarke RM, Jarrett C, Eckersberger E, Levine Z, Schulz WS, Paterson P. Measuring trust in vaccination: A systematic review. Hum Vaccin Immunother. 2018 Jul 3;14(7):1599-1609. doi: 10.1080/21645515.2018.1459252. Epub 2018 May 10. PMID 29617183
- [Background] Karafillakis E, Simas C, Jarrett C, Verger P, Peretti-Watel P, Dib F, De Angelis S, Takacs J, Ali KA, Pastore Celentano L, Larson H. HPV vaccination in a context of public mistrust and uncertainty: a systematic literature review of determinants of HPV vaccine hesitancy in Europe. Hum Vaccin Immunother. 2019;15(7-8):1615-1627. doi: 10.1080/21645515.2018.1564436. Epub 2019 Feb 20. PMID 30633623
- [Background] Holman DM, Benard V, Roland KB, Watson M, Liddon N, Stokley S. Barriers to human papillomavirus vaccination among US adolescents: a systematic review of the literature. JAMA Pediatr. 2014 Jan;168(1):76-82. doi: 10.1001/jamapediatrics.2013.2752. PMID 24276343
- [Background] Fu LY, Bonhomme LA, Cooper SC, Joseph JG, Zimet GD. Educational interventions to increase HPV vaccination acceptance: a systematic review. Vaccine. 2014 Apr 7;32(17):1901-20. doi: 10.1016/j.vaccine.2014.01.091. Epub 2014 Feb 14. PMID 24530401
- [Background] Succi RCM. Vaccine refusal - what we need to know. J Pediatr (Rio J). 2018 Nov-Dec;94(6):574-581. doi: 10.1016/j.jped.2018.01.008. Epub 2018 Apr 12. PMID 29654748
- [Background] Saxena K, Marden JR, Carias C, Bhatti A, Patterson-Lomba O, Gomez-Lievano A, Yao L, Chen YT. Impact of the COVID-19 pandemic on adolescent vaccinations: projected time to reverse deficits in routine adolescent vaccination in the United States. Curr Med Res Opin. 2021 Dec;37(12):2077-2087. doi: 10.1080/03007995.2021.1981842. Epub 2021 Oct 4. PMID 34538163
- [Background] Ryan G, Gilbert PA, Ashida S, Charlton ME, Scherer A, Askelson NM. Challenges to Adolescent HPV Vaccination and Implementation of Evidence-Based Interventions to Promote Vaccine Uptake During the COVID-19 Pandemic: "HPV Is Probably Not at the Top of Our List". Prev Chronic Dis. 2022 Mar 31;19:E15. doi: 10.5888/pcd19.210378. PMID 35358035
- [Background] Patel Murthy B, Zell E, Kirtland K, Jones-Jack N, Harris L, Sprague C, Schultz J, Le Q, Bramer CA, Kuramoto S, Cheng I, Woinarowicz M, Robison S, McHugh A, Schauer S, Gibbs-Scharf L. Impact of the COVID-19 Pandemic on Administration of Selected Routine Childhood and Adolescent Vaccinations - 10 U.S. Jurisdictions, March-September 2020. MMWR Morb Mortal Wkly Rep. 2021 Jun 11;70(23):840-845. doi: 10.15585/mmwr.mm7023a2. PMID 34111058
- [Background] Santoli JM, Lindley MC, DeSilva MB, Kharbanda EO, Daley MF, Galloway L, Gee J, Glover M, Herring B, Kang Y, Lucas P, Noblit C, Tropper J, Vogt T, Weintraub E. Effects of the COVID-19 Pandemic on Routine Pediatric Vaccine Ordering and Administration - United States, 2020. MMWR Morb Mortal Wkly Rep. 2020 May 15;69(19):591-593. doi: 10.15585/mmwr.mm6919e2. PMID 32407298
- [Background] Ateev Mehrotra et al., The Impact of COVID-19 on Outpatient Visits in 2020: Visits Remained Stable, Despite a Late Surge in Cases (Commonwealth Fund, Feb. 2021)
- [Background] Centers for Disease Control and Prevention. Coronavirus Disease 2019 (COVID-19). For Healthcare Professionals. Preserve Supplies. https://www.cdc.gov/coronavirus/2019-ncov/hcp/index.html?CDC_AA_refVal=https%3A%2F%2Fwww.cdc.gov%2Fcoronavirus%2F2019-ncov%2Fhealthcare-facilities%2Findex.html
- [Background] Mann S, Christini K, Chai Y, Chang CP, Hashibe M, Kepka D. Vaccine hesitancy and COVID-19 immunization among rural young adults. Prev Med Rep. 2022 Aug;28:101845. doi: 10.1016/j.pmedr.2022.101845. Epub 2022 Jun 2. PMID 35669235
- [Background] Bar-On YM, Flamholz A, Phillips R, Milo R. SARS-CoV-2 (COVID-19) by the numbers. Elife. 2020 Apr 2;9:e57309. doi: 10.7554/eLife.57309. PMID 32228860
- [Background] Piltch-Loeb R, Silver DR, Kim Y, Norris H, McNeill E, Abramson DM. Determinants of the COVID-19 vaccine hesitancy spectrum. PLoS One. 2022 Jun 1;17(6):e0267734. doi: 10.1371/journal.pone.0267734. eCollection 2022. PMID 35648748
- [Background] Williams CL, Walker TY, Elam-Evans LD, Yankey D, Fredua B, Saraiya M, Stokley S. Factors associated with not receiving HPV vaccine among adolescents by metropolitan statistical area status, United States, National Immunization Survey-Teen, 2016-2017. Hum Vaccin Immunother. 2020 Mar 3;16(3):562-572. doi: 10.1080/21645515.2019.1670036. Epub 2019 Oct 25. PMID 31584312
- [Background] Uva JL, Wagner VL, Gesten FC. Emergency department reliance among rural children in Medicaid in New York State. J Rural Health. 2012 Spring;28(2):152-61. doi: 10.1111/j.1748-0361.2011.00377.x. Epub 2011 Apr 27. PMID 22458316
- [Background] DeGuzman PB, Huang G, Lyons G, Snitzer J, Keim-Malpass J. Rural Disparities in Early Childhood Well Child Visit Attendance. J Pediatr Nurs. 2021 May-Jun;58:76-81. doi: 10.1016/j.pedn.2020.12.005. Epub 2020 Dec 25. PMID 33370620
- [Background] Zablotsky B, Black LI. Prevalence of Children Aged 3-17 Years With Developmental Disabilities, by Urbanicity: United States, 2015-2018. Natl Health Stat Report. 2020 Feb;(139):1-7. PMID 32510313
- [Background] Walker TY, Elam-Evans LD, Yankey D, Markowitz LE, Williams CL, Fredua B, Singleton JA, Stokley S. National, Regional, State, and Selected Local Area Vaccination Coverage Among Adolescents Aged 13-17 Years - United States, 2018. MMWR Morb Mortal Wkly Rep. 2019 Aug 23;68(33):718-723. doi: 10.15585/mmwr.mm6833a2. PMID 31437143
- [Background] Glenn BA, Tsui J, Coronado GD, Fernandez ME, Savas LS, Taylor VM, Bastani R. Understanding HPV vaccination among Latino adolescent girls in three U.S. regions. J Immigr Minor Health. 2015 Feb;17(1):96-103. doi: 10.1007/s10903-014-9996-8. PMID 24557745
- [Background] Mohammed KA, Subramaniam DS, Geneus CJ, Henderson ER, Dean CA, Subramaniam DP, Burroughs TE. Rural-urban differences in human papillomavirus knowledge and awareness among US adults. Prev Med. 2018 Apr;109:39-43. doi: 10.1016/j.ypmed.2018.01.016. Epub 2018 Jan 31. PMID 29378268
- [Background] Shell R, Tudiver F. Barriers to cancer screening by rural Appalachian primary care providers. J Rural Health. 2004 Fall;20(4):368-73. doi: 10.1111/j.1748-0361.2004.tb00051.x. PMID 15551854
- [Background] Peterson CE, Silva A, Holt HK, Balanean A, Goben AH, Dykens JA. Barriers and facilitators to HPV vaccine uptake among US rural populations: a scoping review. Cancer Causes Control. 2020 Sep;31(9):801-814. doi: 10.1007/s10552-020-01323-y. Epub 2020 Jun 14. PMID 32537702
- [Background] Casey MM, Thiede Call K, Klingner JM. Are rural residents less likely to obtain recommended preventive healthcare services? Am J Prev Med. 2001 Oct;21(3):182-8. doi: 10.1016/s0749-3797(01)00349-x. PMID 11567838
- [Background] Yabroff KR, Lawrence WF, King JC, Mangan P, Washington KS, Yi B, Kerner JF, Mandelblatt JS. Geographic disparities in cervical cancer mortality: what are the roles of risk factor prevalence, screening, and use of recommended treatment? J Rural Health. 2005 Spring;21(2):149-57. doi: 10.1111/j.1748-0361.2005.tb00075.x. PMID 15859052
- [Background] Koopman RJ, Mainous AG 3rd, Geesey ME. Rural residence and Hispanic ethnicity: doubly disadvantaged for diabetes? J Rural Health. 2006 Winter;22(1):63-8. doi: 10.1111/j.1748-0361.2006.00009.x. PMID 16441338
- [Background] United States Department of Agriculture. Rural America At a Glance: 2018 Edition. Economic Research Service. Economic Information Bulletin 200. November 2018.
- [Background] Newcomer SR, Freeman RE, Albers AN, Murgel S, Thaker J, Rechlin A, Wehner BK. Missed opportunities for human papillomavirus vaccine series initiation in a large, rural U.S. state. Hum Vaccin Immunother. 2022 Jan 31;18(1):2016304. doi: 10.1080/21645515.2021.2016304. Epub 2022 Feb 4. PMID 35119342
- [Background] Centers for Disease Control and Prevention. Human Papillomavirus (HPV). Cancers Caused by HPV. . Available from: https://www.cdc.gov/hpv/parents/cancer.html
- [Background] Kepka D, Spigarelli MG, Warner EL, Yoneoka Y, McConnell N, Balch A. Statewide analysis of missed opportunities for human papillomavirus vaccination using vaccine registry data. Papillomavirus Res. 2016 Dec;2:128-132. doi: 10.1016/j.pvr.2016.06.002. PMID 27540595
- [Background] Centers for Disease Control and Prevention. HPV-Associated Cancers Rates by Race and Ethnicity. 2019. Atlanta
- [Background] Bruno DM, Wilson TE, Gany F, Aragones A. Identifying human papillomavirus vaccination practices among primary care providers of minority, low-income and immigrant patient populations. Vaccine. 2014 Jul 16;32(33):4149-54. doi: 10.1016/j.vaccine.2014.05.058. Epub 2014 Jun 2. PMID 24886959
- [Background] Katz ML, Reiter PL, Heaner S, Ruffin MT, Post DM, Paskett ED. Acceptance of the HPV vaccine among women, parents, community leaders, and healthcare providers in Ohio Appalachia. Vaccine. 2009 Jun 19;27(30):3945-52. doi: 10.1016/j.vaccine.2009.04.040. Epub 2009 May 3. PMID 19389447
- [Background] Vanderpool RC, Dressler EV, Stradtman LR, Crosby RA. Fatalistic beliefs and completion of the HPV vaccination series among a sample of young Appalachian Kentucky women. J Rural Health. 2015 Spring;31(2):199-205. doi: 10.1111/jrh.12102. Epub 2015 Jan 14. PMID 25640763
- [Background] Blumling AA, Thomas TL, Stephens DP. Researching and Respecting the Intricacies of Isolated Communities. Online J Rural Nurs Health Care. 2013;13(2):Blumling. PMID 24817833
- [Background] Head KJ, Vanderpool RC, Mills LA. Health care providers' perspectives on low HPV vaccine uptake and adherence in Appalachian Kentucky. Public Health Nurs. 2013 Jul;30(4):351-60. doi: 10.1111/phn.12044. Epub 2013 Apr 8. PMID 23808860
- [Background] Henley SJ, Anderson RN, Thomas CC, Massetti GM, Peaker B, Richardson LC. Invasive Cancer Incidence, 2004-2013, and Deaths, 2006-2015, in Nonmetropolitan and Metropolitan Counties - United States. MMWR Surveill Summ. 2017 Jul 7;66(14):1-13. doi: 10.15585/mmwr.ss6614a1. PMID 28683054
- [Background] Centers for Disease Control and Prevention. TeenVaxView. Vaccination Coverage among Adolescents (13 - 17 Years). . Available from: https://www.cdc.gov/vaccines/imz-managers/coverage/teenvaxview/data-reports/index.html
- [Background] U.S. Department of Health and Human Services. Office of Disease Prevention and Health Promotion. Healthy People 2030. Increase the proportion of adolescents who get recommended doses of the HPV vaccine - IID-08. Available from: https://health.gov/healthypeople/objectives-and-data/browse-objectives/vaccination/increase-proportion-adolescents-who-get-recommended-doses-hpv-vaccine-iid-08.
- [Background] Centers for Disease Control and Prevention. How Many Cancers Are Linked with HPV Each Year? Available from: https://www.cdc.gov/cancer/hpv/statistics/cases.htm.
- See also: PREVENT HPV Cancers study website hosted by Kaiser Permanente — https://preventhpvcancers.com/
- See also: PREVENT HPV Cancers study website hosted by Kaiser Permanente — https://research.kpchr.org/preventhpvcancers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | English Language Session and Messaging | Spanish Language Session and Messaging
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | English Language Session and Messaging | Spanish Language Session and Messaging | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.13 (7.43) | 40.50 (7.06) | 41.67 (7.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 4 | 1 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 8 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18
Likelihood of Parents to Get the HPV Vaccination for Their Child(ren) This Year [Count of Participants; unit: Participants] — Participants will be surveyed before and after the in-person session to assess learning outcomes.
  This outcome measure is a single-item self-report of the intention of parents to get the HPV vaccination for their children this year. A low score (Minimum: 1 Extremely Unlikely) is an unfavorable outcome and a high score (Maximum: 5 Extremely Likely) is a favorable outcome. This outcome measure will report the number of patients per response for the BCT English sessions and the BCT Spanish sessions.
  Participants
    Extremely likely | 3 | 0 | 3
    Likely | 1 | 3 | 4
    Neutral | 2 | 1 | 3
    Unlikely | 1 | 1 | 2
    Extremely unlikely | 0 | 0 | 0
    My child(ren) has already received the HPV vaccine | 1 | 1 | 2
    Prefer not to answer | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Parents Participating in BCT
Description: This outcome measure will report the number of participants who participant in the BCT English sessions and number of participants who participant in the BCT Spanish sessions.
  BCT is a community-based research approach to develop and evaluate messaging for health related issues. This study will employ BCT to determine the frequency and content of HPV messaging for future research.
Time Frame: 1 day after study enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | English Language Session and Messaging | Spanish Language Session and Messaging
Number analyzed (Participants) | 8 | 10
Participants | 8 | 10

2. Secondary Outcome: Likelihood of Parents to Get the HPV Vaccination for Their Child(Ren) This Year
Description: Participants will be surveyed before and after the in-person session to assess learning outcomes.
  This outcome measure is a single-item self-report of the intention of parents to get the HPV vaccination for their children this year. A low score (Minimum: 1 Extremely Unlikely) is an unfavorable outcome and a high score (Maximum: 5 Extremely Likely) is a favorable outcome. This outcome measure will report the number of patients per response for the BCT English sessions and the BCT Spanish sessions.
Time Frame: After the in-person session (1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | English Language Session and Messaging | Spanish Language Session and Messaging
Number analyzed (Participants) | 8 | 10
Participants
  Extremely likely | 6 | 1
  Likely | 1 | 5
  Neutral | 0 | 1
  Unlikely | 0 | 0
  Extremely unlikely | 0 | 2
  My child(ren) has already received the HPV vaccine | 1 | 1
  Prefer not to answer | 0 | 0

3. Secondary Outcome: Satisfaction With BCT Session
Description: Participants will be surveyed before and after the in-person session to assess learning outcomes.
  This outcome measure is a single-item self-report of the participants satisfaction with the BCT session. A low score (Minimum: 1 Not at all satisfied) is an unfavorable outcome and a high score (Maximum: 10 Extremely satisfied) is a favorable outcome. This outcome measure will report the mean score of participants for the BCT English sessions and the BCT Spanish sessions.
Time Frame: After the in-person session (1 day)
Population: One participant in the English Language Session did not answer this item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | English Language Session and Messaging | Spanish Language Session and Messaging
Number analyzed (Participants) | 7 | 10
units on a scale | 9.71 (0.49) | 9.10 (1.29)

ADVERSE EVENTS:
Time Frame: Adverse event data was not collected for this study.
Description: Adverse event data was not collected for this study.
Arm/Group | English Language Session and Messaging | Spanish Language Session and Messaging
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT06290206/Prot_SAP_000.pdf